CLINICAL TRIAL: NCT00898469
Title: Study Of Pharmacogenetic Risk Factors For Avascular Necrosis CCG 1882
Brief Title: Identifying Risk Factors for Bone Tissue Death in Young Patients With Acute Lymphoblastic Leukemia Treated on Clinical Trial CCG-1882
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL03B2; COG-AALL03B2 (Other: Children's Oncology Group); CDR0000304752 (Other: Clinical Trials.gov)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: polymorphism analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to bone tissue death.

PURPOSE: This laboratory study is looking at risk factors for bone tissue death in young patients with acute lymphoblastic leukemia treated on clinical trial CCG-1882.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify possible pharmacogenetic risk factors for avascular necrosis (AVN) in pediatric patients who received intensive therapy for acute lymphoblastic leukemia on clinical trial CCG-1882.
* Compare whether thymidylate synthase 2/2 enhancer repeat genotype and vitamin D receptor C/C start site genotype are more common among patients who developed AVN than among patients who did not.

OUTLINE: This is a retrospective, cohort, multicenter study. Patients are stratified according to gender and treatment regimen on clinical trial CCG-1882 (augmented vs regular Berlin-Frankfurt-Munster).

DNA is extracted from slides of blast samples that were previously obtained from patients treated on clinical trial CCG-1882. DNA genotyping is performed, and genotypes (proportion of population with variant alleles or frequency of variant alleles) are compared between patients who did and did not develop avascular necrosis.

PROJECTED ACCRUAL: A total of 671 tissue samples from patients (294 females and 377 males) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia (ALL)

  * Has diagnostic ALL blast sample slides available for DNA extraction
* Previously treated on clinical trial CCG-1882

PATIENT CHARACTERISTICS:

Age

* 10 and over at diagnosis

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 10 Years to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients who received intensive therapy for acute lymphoblastic leukemia on clinical trial CCG-1882.
Sampling Method: Non-Probability Sample
Enrollment: 671 (Estimated)
Dates: Start 2005-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Identification of possible pharmacogenetic risk factors for avascular necrosis | length of study
Comparison of whether thymidylate synthase 2/2 enhancer repeat genotype and vitamin D receptor C/C start site genotype are more common among patients who developed avascular necrosis than among patients who did not | length of study

CONTACTS AND LOCATIONS:
Overall Officials: Mary Relling, PharmD, Study Chair — St. Jude Children's Research Hospital

REFERENCES:
- [Result] Hamilton LH, Mattano LA, Sather HN, et al.: A SERPINE1 (PAI-1) single nucleotide polymorphism predicts osteonecrosis in children treated for acute lymphoblastic leukemia: results of the Childrens Oncology Group (COG) study AALL03B2. [Abstract] Blood 108 (11): A-709, 2006.